CLINICAL TRIAL: NCT04880512
Title: A Double-blinded, Randomized, Placebo-controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SYHX1901 Tablets in Chinese Healthy Subjects
Brief Title: The Safety, Tolerability, and Pharmacokinetics of SYHX1901 Tablets in Chinese Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYHX1902-CSP-001
Record Dates: First submitted 2021-04-27; First posted 2021-05-10 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SYHX 1901 tablets for SAD (Experimental): Two subjects will be enrolled in a single dose group which is recommended as the initial dose. 8 out of 10 healthy subjects will be randomized to receive a single dose of SYHX 1901 tablets in fasted state.
  Interventions: Drug: SYHX 1901 tablets
- Placebo for SAD (Placebo Comparator): 2 out of 10 healthy subjects will be randomized to receive a single dose of placebo in fasted state
  Interventions: Drug: Placebo
- SYHX 1901 tablets for MAD (Experimental): 8 out of 10 healthy subjects will be randomized to receive multiple doses of SYHX 1901 tablets in fasted state
  Interventions: Drug: SYHX 1901 tablets
- Placebo for MAD (Placebo Comparator): 2 out of 10 healthy subjects will be randomized to receive multiple doses of placebo in fasted state
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYHX 1901 tablets — SYHX 1901, oral tablets, in fasted state
  Arms: SYHX 1901 tablets for MAD; SYHX 1901 tablets for SAD
Drug: Placebo — Matching placebo, oral tablets, in fasted state
  Arms: Placebo for MAD; Placebo for SAD

SUMMARY:
This is a phase I clinical trial to evaluate the safety, tolerability and pharmacokinetic characteristics of single ascending doses and multiple ascending doses of SYHX1901 tablets in Chinese healthy subjects

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and pharmacokinetic characteristics of single ascending doses (part 1) and multiple ascending doses (part 2) of SYHX1901 tablets in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 45 years (inclusive)；
2. Have a body mass index (BMI) between 18.0 and 26.0 kg/m2 (inclusive) and weigh at least 45.0 kg (female) or 50.0 kg (male) at screening；
3. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, vital signs, physical examination, and clinical laboratory tests (hematology, urinalysis, and coagulation)；
4. Subjects and their partners agree to use effective n4. Subjects and their partners agree to use effective non-hormonal contraceptive measures (e.g., condoms, inert intrauterine devices, female barriers (cervix cap or diaphragm with spermicide), vaginal contraceptive ring, etc.) from signing the informed consent form to 6 months after the end of the study, or have taken permanent contraceptive measures (e.g., bilateral fallopian tube ligation, vasectomy, etc.); male subjects have no sperm donation plan from signing the informed consent to 6 months after the end of the study, female subjects have no egg donation plan from signing the informed consent form to 6 months after the end of the study；
5. Subjects who fully understand the study, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Prior neurological/ psychiatric, respiratory system, endocrine system, blood system, skeletal-muscular system diseases or liver and kidney dysfunction or other diseases that may affect the results of the study;
2. History of severe allergies, herpes zoster infection, or tuberculosis;
3. Those who have taken any prescription drugs, over-the-counter drugs, proprietary Chinese medicines, herbal medicines, vitamin dietary supplements and health products within 4 weeks before signing the informed consent, and those who use oral long-acting contraceptives or use embedded long-acting contraceptives；
4. Subjects with diseases affecting drug absorption, distribution, metabolism and excretion as judged by investigator (e.g., acute and chronic diarrhea, acute and chronic gastritis, etc.);
5. Surgery history within 6 months prior to signing the informed consent;
6. Subjects with surgery plan (including cosmetic surgery, dental surgery and oral surgery), or strenuous exercise plan (including physical contact sports or collision sports) during the trial period;
7. Subjects with any clinically significant abnormalities in ECG, QTcF interval greater than 450 ms (male) or 470 ms (female), or with a history of prolonged QTcF interval;
8. Subjects with one or more abnormalities in the vital signs at screening: ear temperature >37.5ºC, pulse rate >100 beats/min, systolic blood pressure ≥140 mmHg or <90 mmHg, diastolic blood pressure >90 mmHg or <50 mmHg；
9. The white blood cell count, the absolute value of neutrophils and the absolute value of lymphocytes are below the lower limit or higher than the upper limit of the reference value, and the percentage of reticulocyte (RET) is below the lower limit of the reference value in routine blood tests at screening;
10. History of acute respiratory or systemic infections within 2 weeks before signing the informed consent;
11. Blood lost or donation more than 400 mL within 3 months before signing the informed consent;
12. Alcohol abuse: consumption of more than 14 units of alcohol per week within 4 weeks prior to signing the informed consent or positive test for Alcohol at screening；
13. Smoker: more than 5 cigarettes per day within 6 months prior to signing informed consent；
14. Habitual intake of excessive xanthine- or caffeine-containing food, beverages, or other factors, which may interfere the absorption, distribution, metabolism, or excretion of drugs, within 4 weeks prior to screening；
15. Subjects have participated in clinical trials of any drug or medical device within 3 months before signing the informed consent;
16. History of substance abuse within the 1 years prior to signing the informed consent, or positive test for drug abuse at screening；
17. Female subjects who are pregnant or lactating;
18. Anti-Mullerian hormone (female only) test results not within the reference range at screening;
19. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (anti-HCV), Human immunodeficiency virus antibody (anti-HIV) or Treponema Pallidum antibody (Anti-TP) at screening；
20. Suspected or known allergy to the test drug or any ingredient in the test drug, or subjects with allergic constitution;
21. Not suitable for this trial as determined by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SYHX1901 tablets | SAD: up to14 days after the dosing, MAD: up to 7 days after the last dosing
  The safety and tolerability of single or multiple doses of SYHX1901 tablets administered orally will be assessed by incidence and severity of adverse events (AEs), abnormalities in clinical laboratory assessments, ECGs, vital sign assessments, and physical exams.

SECONDARY OUTCOMES:
The PK of SYHX1901 following single-dose and multiple doses | Pre-dose and multiple timepoints up to 144 hours after the last dose
  Peak Plasma Concentration (Cmax) of SYHX1901 following single-dose and multiple doses
The PK of SYHX1901 following single-dose and multiple doses | Pre-dose and multiple timepoints up to 144 hours after the last dose
  Area under the plasma concentration versus time curve (AUC) of SYHX1901 following single-dose and multiple doses
The PK of SYHX1901 following single-dose and multiple doses | Pre-dose and multiple timepoints up to 144 hours after the last dose
  The concentration peak time of SYHX1901 following single-dose and multiple doses
  Concentration peak time
  The peak time of SYHX1901 concentration following single-dose
The PK of SYHX1901 following single-dose and multiple doses | Pre-dose and multiple timepoints up to 144 hours after the last dose
  The half-time of SYHX1901 following single-dose and multiple doses
  The half - time of SYHX1901 following single-dose
The PK of SYHX1901 following single-dose and multiple doses | Pre-dose and multiple timepoints up to 144 hours after the last dose
  The plasma clearance rate （CL）of SYHX1901 following single-dose and multiple doses
Urine PK parameters | Pre-dose and multiple timepoints up to 144 hours after the dose（180 mg）
  Urine pharmacokinetic parameters: The Urine clearance rate （CLr）of SYHX1901
Urine PK parameters | Pre-dose and multiple timepoints up to 144 hours after the dose（180 mg）
  Urine pharmacokinetic parameters: Cumulative excretion from time t1 to t2(Aet1-t2)
  Fecal pharmacokinetic parameters:Cumulative excretion from time t1 to t2
  Urine pharmacokinetic parameters:cumulative excretion from time t1 to t2
Fecal PK parameters | Pre-dose and multiple timepoints up to 144 hours after the dose（180 mg）
  Fecal pharmacokinetic parameters: cumulative excretion from time t1 to t2(Aft1-t2)
Identification of Metabolites of SYHX1901 | Pre-dose and multiple timepoints up to 144 hours after the dose（180 mg）
  It is a prospective study aiming to characterize metabolites of 1901 in human plasma, urine and feces. The metabolism profiles of 1901 and main metabolites will be build up.
PD indexes: the level of PSTATs in blood cells | Pre-dose and multiple timepoints up to 144 hours after the last dose
  Pharmacodynamic indexes: the level of PSTATs in blood cells
PD indexes: the inhibition rate of PSTATs in blood cells | Pre-dose and multiple timepoints up to 144 hours after the last dose
  Pharmacodynamic indexes: the inhibition rate of PSTATs in blood cells

CONTACTS AND LOCATIONS:
Overall Officials: jing zhang, Medical PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, China